CLINICAL TRIAL: NCT00061217
Title: Comparison of Rectified and Unrectified Amputee Sockets
Brief Title: Prosthetic Limbs After Leg Amputation: Alternative Method of Socket Design
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R01HD038919-02 (NIH)
Record Dates: First submitted 2003-05-22; First posted 2003-05-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-10

CONDITIONS: Amputation
Keywords: Transtibial amputees; Rectified sockets; Unrectified sockets; Gait; Energy expenditure; Prosthetic evaluation questionnaire

INTERVENTIONS:
Device: Unrectified prosthetic socket
Device: Rectified prosthetic socket

SUMMARY:
People who have had a leg amputated often choose to use a prosthetic (artificial) leg. This study will evaluate a new method of making prosthetic legs for people who have had an amputation below the knee.

DETAILED DESCRIPTION:
The traditional assumption when fabricating a transtibial amputee (TTA) socket is that the residual limb is not homogeneous in its ability to tolerate load. As a result, prosthetic sockets are currently fabricated by modifying a positive mold to account for this non-homogeneity; these are called rectified sockets. Unrectified sockets retain the shape of the residual limb, except for a distal end pad. Unrectified sockets use an alginate gel method of fabricating that is simpler and less time consuming than the method used to fabricate rectified sockets. This study will compare patient satisfaction and function with rectified and unrectified sockets.

Participants in this study will be randomized to either a recitified socket group or an unrectified socket group. Participants will wear the socket for a minimum of 4 weeks. Participants will then fill out a Prosthesis Evaluation Questionnaire (PEQ). The PEQ quantifies patient satisfaction by evaluating nine validated scales. Functional measures of energy expenditure, kinematics, and ground reaction forces during gait will also be collected. After 4 weeks, participants in the rectified socket group will switch to an unrectified socket and participants in the unrectified socket group will switch to a rectified socket. At the end of 4 weeks with the new socket, participants will once again fill out the PEQ and undergo functional assessment. At the end of study participation, each participant will freely choose the socket they wish to have in their final prosthesis.

Thus far, 10 study participants with unilateral transtibial amputations have been evaluated after randomly wearing both rectified and unrectified sockets for 4 weeks. Results indicated no differences between sockets for gait speed and timing, gait kinematics and kinetics, gait energy expenditure, and Rate of Perceived Exertion (RPE). There were also no differences in the Prosthetic Evaluation Questionnaire. Four participants selected the rectified socket and 6 selected the unrectified socket as their exit socket.

ELIGIBILITY:
Inclusion Criteria

* Unilateral transtibial amputation
* Mature residual limbs (i.e., no major change in stump volume due to atrophy or other destabilizing factors)
* Continuously worn a prosthesis for at least 1 year prior to study entry
* Scheduled for a new prosthesis
* Independent ambulation
* No acute health problems

Exclusion Criteria

* Constant recurring prosthetic problems (i.e., adherent scar tissue, neuromas, bony protuberances at distal end)
* Requires gel inserts, additional ply socks, or other atypical fitting components or methods
* Health status that prohibits patient from performing graded exercise test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59
Dates: Start 2001-04; Study Completion 2005-03

PRIMARY OUTCOMES:
socket selection
PEQ
gait speed

SECONDARY OUTCOMES:
gait kinematics
gait kinetics
energy consumption

CONTACTS AND LOCATIONS:
Overall Officials: Jack R. Engsberg, Ph.D., Principal Investigator
Locations (1):
- Jack R. Engsberg, St Louis, Missouri, United States

REFERENCES:
- [Background] Engsberg JR, Sprouse SW, Uhrich ML, Ziegler BR, Luitjohan FD. Comparison of Rectified and Unrectified Sockets for Transtibial Amputees. J Prosthet Orthot. 2008;18(1):1-7. doi: 10.1097/00008526-200601000-00002. PMID 18776945